CLINICAL TRIAL: NCT07028099
Title: Multi-Center Randomized Controlled Clinical Study on the Application of a Novel Expandable Posterior Bone Grafting OLIF Cage
Brief Title: A Study on the Clinical Use of a New Expandable OLIF Cage With Posterior Bone Grafting in Lumbar Spine Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Peking University People's Hospital (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Jinan Hospital, Xuanwu Hospital, Capital Medical University (Unknown); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Shanghai changzheng hospital, Naval Medical University (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QYFYEC2025-62
Record Dates: First submitted 2025-06-10; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Spondylolisthesis; Degenerative Lumbar Scoliosis; Lumbar Disc Herniation; Lumbar Spinal Stenosis
Keywords: Expandable OLIF Cage; Minimally Invasive Spine Surgery; Prospective Multicenter Randomized Controlled Trial; Degenerative Lumbar Disease
MeSH Terms: conditions — Spondylolisthesis; Intervertebral Disc Displacement; Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (Active Comparator)
  Interventions: Device: Conventional OLIF cage
- Experimental group (Experimental)
  Interventions: Device: Expandable OLIF cage with posterior bone grafting

INTERVENTIONS:
Device: Expandable OLIF cage with posterior bone grafting — This intervention involves the use of a novel expandable OLIF cage that allows intraoperative height adjustment and posterior bone grafting through a dedicated channel. The device is designed to restore intervertebral height and lumbar lordosis while minimizing endplate injury. Bone grafts (autologous or synthetic) are delivered after expansion to enhance fusion. This design aims to reduce cage subsidence, improve fusion rates, and simplify the surgical workflow compared to conventional OLIF cages with fixed heights.
  Arms: Experimental group
Device: Conventional OLIF cage — Participants in the control group will undergo oblique lateral interbody fusion (OLIF) using a standard non-expandable interbody fusion cage. The cage has a fixed height and is inserted via the retroperitoneal approach. Bone grafts are packed into the cage prior to insertion through the anterior or lateral window. This represents the current standard practice for OLIF procedures and does not allow intraoperative height adjustment or posterior graft delivery. The procedure follows conventional OLIF surgical protocols without additional design modifications.
  Arms: Control group

SUMMARY:
This clinical trial aims to evaluate the safety and effectiveness of a novel expandable OLIF (Oblique Lateral Interbody Fusion) cage with posterior bone grafting in patients with lumbar degenerative diseases. OLIF is a minimally invasive spinal surgery technique that restores intervertebral height and relieves nerve compression by placing a cage into the disc space.

The new device allows surgeons to adjust the height of the cage during surgery and deliver bone grafts through a special channel after expansion. This study compares the outcomes of patients receiving the new cage versus those treated with a conventional OLIF cage.

The trial will assess pain relief, functional improvement, spinal stability, fusion success, and potential complications. Radiological images and patient-reported scores (like VAS and ODI) will be collected over 12 months. The study includes patients aged 40 to 80 with single-level lumbar spine disease who have not improved after at least 6 months of conservative treatment.

This study will help determine whether the new expandable cage offers clinical advantages and better long-term outcomes for patients undergoing OLIF surgery.

ELIGIBILITY:
Inclusion Criteria:1: Age between 40 and 80 years (inclusive)

2: Clinically diagnosed with lumbar spondylolisthesis or lumbar spinal stenosis

3: Confirmed single-level lumbar degenerative disease

4: Affected level located at L2/3, L3/4, or L4/5

5: Failure of conservative treatment for at least 6 months

Exclusion Criteria:1: Patients requiring direct decompression of the spinal canal

2: History of prior lumbar or retroperitoneal surgery

3: Abnormal anatomy between the iliac vascular sheath and the psoas major muscle

4: Presence of active infection or other significant systemic diseases

5: Inability to complete surgical treatment or comply with follow-up due to various limitations

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative cage subsidence | From enrollment to the 12th month after operation
  Radiological follow-up will be conducted immediately after surgery, and at 6, 12 months postoperatively using X-ray and/or CT imaging. Cage subsidence is defined as: ≥2 mm of cage penetration into the adjacent vertebral endplate compared to immediate postoperative imaging; Visible collapse of the cage-endplate interface; ≥10% reduction in intervertebral height compared to initial postoperative height. All radiographic assessments will be performed independently by two spine surgeons or radiologists blinded to group allocation. In case of discrepancy, a third reviewer will adjudicat
ntraoperative cartilage endplate injury | From enrollment to the 12th month after operation
  Endplate injury will be assessed intraoperatively by the operating surgeon through direct visual inspection and intraoperative fluoroscopy. Injury is defined as any of the following: Visible collapse, fracture, or tearing of the cartilaginous endplate during cage insertion; Evidence of asymmetric or excessive endplate compression on fluoroscopy; Explicit documentation of "endplate injury" or "endplate violation" in the operative record. Injury will be recorded in binary form (Yes/No). When necessary, postoperative CT scans may be used to confirm suspected endplate damage.

SECONDARY OUTCOMES:
Intervertebral Height | From enrollment to the 12th month after operation
  On lateral X-ray or CT images, the target intervertebral space is selected, and the intervertebral space heights of the leading edge, middle point and trailing edge are measured respectively, and the average value is taken to represent the intervertebral height of this segment.
Clinical efficacy index of patients: VAS | From enrollment to the 12th month after operation
  Visual Analog Scale, (VAS) of pain. Measurement method: Patients were evaluated by VAS score before operation, 3 months, 6 months and 12 months after operation. Use a horizontal scale of 10 cm, with one end marked as "0 = painless" and the other end marked as "10 = the most severe pain". The patient draws a line on the ruler according to his own feelings, and measures the distance (in centimeters) from the starting point of "0" to the drawing point as the scoring result..
Cobb angle of lumbar coronal plane | From enrollment to the 12th month after operation
  Used to evaluate lumbar scoliosis or coronal imbalance. Measurements are performed on preoperative and postoperative standing anteroposterior (AP) lumbar spine radiographs or coronal CT reconstructions. Identify the most tilted upper end vertebra and the most tilted lower end vertebra in the coronal plane; Draw lines along the upper endplate of the upper vertebra and the lower endplate of the lower vertebra; Construct perpendicular lines to each endplate line; The angle between these two perpendiculars is recorded as the coronal Cobb angle. The angle is recorded in degrees (°).
Cobb angle of lumbar deformity surface | From enrollment to the 12th month after operation
  Draw lines along the superior endplate of L1 and the superior endplate of S1; The angle formed between these two lines is defined as the sagittal Cobb angle (lumbar lordosis angle). The angle is recorded in degrees (°).
Clinical efficacy index of patients: ODI | From enrollment to the 12th month after operation
  Oswestry Disability Index, (ODI). Measurement method: The Chinese version of ODI scale was used, which was completed by patients' self-evaluation, including 10 items (such as pain intensity, personal care, walking, social life, etc.), and each item was scored at 5 levels. The total score is 50 points.In this study, a lower ODI score postoperatively reflects better functional recovery and greater treatment effectiveness.

IPD SHARING:
Plan to Share IPD: Yes
The individual participant data (IPD) underlying the results of this study will be available upon reasonable request from qualified researchers. Access will be granted after the approval of a data-sharing agreement and ethical clearance. De-identified datasets will be provided to ensure patient confidentiality.

DOCUMENTS (2):
  • Study Protocol (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT07028099/Prot_000.pdf
  • Informed Consent Form (2025-04-21): https://cdn.clinicaltrials.gov/large-docs/99/NCT07028099/ICF_001.pdf